CLINICAL TRIAL: NCT01294605
Title: Double-blind, Randomized, Phase III Clinical Trial to Evaluate the Immunogenicity and Reactogenicity of Three Consecutive Doses of dTpa, or of dTpa-IPV Followed by Two Doses of Td Vaccine , and Compared to Three Consecutive Doses of Td Vaccine Administered to Healthy Adults in a 0,1,6-month Schedule
Brief Title: Immunogenicity and Reactogenicity Study of BoostrixTM (dTpa) and Boostrix-IPV (dTpa-IPV)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 263855/034
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Acellular Pertussis; Tetanus; Diphtheria
Keywords: DTPa; Td; IPV
MeSH Terms: conditions — Tetanus; Diphtheria | interventions — Boostrix; Pentetic Acid; Tetanus Toxoid; Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Group A (Experimental)
  Interventions: Biological: Boostrix™ (dTpa)
- Group B (Experimental)
  Interventions: Biological: GSK Biologicals' reduced-antigen-content combined diphtheria, tetanus, acellular pertussis and inactivated polio vaccine (dTpa-IPV; BoostrixTM); Biological: Ditanrix™ Adult, TedivaxTM (Td)
- Group C (Active Comparator)
  Interventions: Biological: Ditanrix™ Adult, TedivaxTM (Td)

INTERVENTIONS:
Biological: Boostrix™ (dTpa) — Intramuscular, 3 doses
  Arms: Group A
Biological: GSK Biologicals' reduced-antigen-content combined diphtheria, tetanus, acellular pertussis and inactivated polio vaccine (dTpa-IPV; BoostrixTM) — Intramuscular, single dose
  Arms: Group B
Biological: Ditanrix™ Adult, TedivaxTM (Td) — Intramuscular, 2 doses
  Arms: Group B
Biological: Ditanrix™ Adult, TedivaxTM (Td) — Intramuscular, 3 doses
  Arms: Group C

SUMMARY:
This purpose of the study is to evaluate the immunogenicity and reactogenicity of Boostrix™ (when used in a primary schedule (0, 1, 6-month) or a single dose of Boostrix-IPV followed by two doses of Td vaccines (DitanrixTM Adult, TedivaxTM), as compared to three doses of licensed Td vaccines in adults.

ELIGIBILITY:
Inclusion Criteria:

* Only subjects for whom the investigator believes the requirements of the protocol will be complied with will be enrolled in the study
* A male or female adult >= 40 years of age
* Written informed consent to be obtained from the subject prior to study entry
* No history of diphtheria or tetanus toxoid containing vaccination in the last 20 years, including those who have never been vaccinated and those with an unknown vaccination status.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* subject should not be pregnant or plan to become pregnant.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* Pregnant or lactating female
* Female planning to become pregnant or planning to discontinue contraceptive precautions
* Previous vaccination with a meningococcal-conjugate vaccine, Prevenar™ or other experimental conjugated pneumococcal vaccines
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine(s).
* Any confirmed or suspected immunosuppressive or immunodeficient condition

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2003-04; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Immunogenicity with respect to components of the study vaccines | One month after the third dose (Month 7)

SECONDARY OUTCOMES:
Immunogenicity with respect to components of the study vaccines | One month after each dose (Months 1, 2 and 7)
Occurrence of solicited local and general symptoms | Within 15 days (day 0 -14) after each vaccine dose.
Occurrence of unsolicited symptoms | Within 31 days (day 0-30) after each vaccine dose.
Occurrence of serious adverse events | Until 31 days (day 0-30) after the last vaccine dose.
Occurrence of large local swelling reported | Within 15 days (day 0-14) after each vaccine dose
Use of concomitant medication taken | Within 31 days (day 0-30) after each vaccine dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- Belgium (3):
  - GSK Investigational Site, Bruges
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Wilrijk
- Netherlands (2):
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Utrecht
- Spain (6):
  - GSK Investigational Site, Alzira
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Centelles
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Mollet del Vallès
  - GSK Investigational Site, Vic

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Theeten H, Rumke H, Hoppener FJ, Vilatimo R, Narejos S, Van Damme P, Hoet B. Primary vaccination of adults with reduced antigen-content diphtheria-tetanus-acellular pertussis or dTpa-inactivated poliovirus vaccines compared to diphtheria-tetanus-toxoid vaccines. Curr Med Res Opin. 2007 Nov;23(11):2729-39. doi: 10.1185/03007x233034. PMID 17897485
- [Background] Van Damme P, McIntyre P, Grimprel E, Kuriyakose S, Jacquet JM, Hardt K, Messier M, Van Der Meeren O. Immunogenicity of the reduced-antigen-content dTpa vaccine (Boostrix((R))) in adults 55 years of age and over: a sub-analysis of four trials. Vaccine. 2011 Aug 11;29(35):5932-9. doi: 10.1016/j.vaccine.2011.06.049. Epub 2011 Jun 28. PMID 21718738
- [Background] Van Damme P et al. Primary vaccination of adults with reduced antigen content diphtheria-tetanus-acellular pertussis (dTpa) vaccines. Abstract presented at the 27th Annual Meeting of European Society for Paediatric Infectious Diseases (ESPID), Brussels, Belgium. 09-13 June 2009.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 263855/034 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 263855/034 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 263855/034 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 263855/034 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 263855/034 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 263855/034 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register